CLINICAL TRIAL: NCT04452136
Title: 68Ga PSMA-11 in Patients With Intermediate to High-risk Prostate Cancer Before Prostatectomy or With Biochemical Recurrence of Prostate Cancer.
Brief Title: Expanded Access Protocol of 68Ga PSMA 11 PET Imaging of Prostate Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Jeanne Link (Other)
Collaborators: OHSU Center of Radiochemistry Research (Unknown); Oregon Health and Science University (Other); OHSU Knight Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Jeanne Link, Professor, OHSU Knight Cancer Institute
Organization: OHSU Knight Cancer Institute (Other)
Other Study IDs: STUDY00020072; STUDY00020073 (Other: OHSU Knight Cancer Institute IRB Number)
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Prostatic Neoplasms; Prostatic Diseases; Prostate Cancer; Prostate Cancer Metastatic; Prostate Cancer Recurrent
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: 68GA PSMA-HBED-CC — Given IV
  Other Names: 68Ga-PSMA-11

SUMMARY:
This study provides expanded access to radiotracer Gallium 68 (68Ga)-prostate-specific membrane antigen (PSMA)-HBED-CC (68Ga-PSMA-11) with Positron Emission Tomography (PET) imaging for participants with intermediate and high risk prostate cancer before prostatectomy or for suspected biochemical recurrence of their prostate cancer. Compared to conventional imaging, 68Ga PSMA-HBED-CC might improve the ability to localize the sites of recurrent or metastatic disease, which helps with surgical and other treatment planning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Provide participants with prostate cancer access to 68Ga PSMA-HBED-CC to localize the site of potential metastatic or recurrent disease.

OUTLINE:

Eligible participants will be intravenously administered 68Ga PSMA-HBED-CC at a dose of 3-7 mCi (111 - 259 MBq), target 5 mCi. The estimated uptake time of the study agent is 75 minutes ± 25 minutes. The targeted uptake time is 60 minutes, with an acceptable range of 50-100 minutes. Following the PET scan with the study agent, participants will undergo either surgical management or treatment for metastatic disease in accordance with institutional standards.

Patients will be observed for 2 hours after injection of the radiotracer, and will be followed-up 1-3 days post injection with a phone call.

ELIGIBILITY:
Inclusion Criteria:

PLANNED PROSTATECTOMY

* Biopsy-proven prostate adenocarcinoma
* Intermediate to high-risk disease, defined as one of the following factors: PSA > 10, T2b or greater, or a Gleason score of 7 or greater.
* Planned prostatectomy with lymph node dissection
* Must be treatment naïve (not have received neoadjuvant chemotherapy, radiation therapy, hormonal therapy, androgen deprivation therapy, or focal ablation techniques (e.g., HiFu)

BIOCHEMICAL RECURRENCE

* Pathologically proven prostate adenocarcinoma. Rising PSA after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy).
* If post-radical prostatectomy, PSA > 0.2 ng/mL measured > 6 weeks post-operatively and confirmatory persistent PSA greater than 0.2 ng/mL (AUA recommendation for biochemical recurrence).
* If post-radiation therapy, PSA that is equal to or greater than a 2 mg/mL rise above PSA nadir (ASTRO recommendation for biochemical recurrence).
* No other malignancy within the past 2 years (skin basal cell or cutaneous superficial squamous cell carcinoma or superficial bladder cancer are exempt from this criterion).

ALL

* Karnofsky performance status (KPS) >= 50 (ECOG/WHO 0, 1, or 2)
* Not receiving any other investigational agents (i.e., unlabeled drugs or drugs under an IND for initial efficacy investigations
* Ability to understand and the willingness to provide informed consent

Exclusion Criteria:

* History of Stevens-Johnson syndrome
* Known Paget's disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Mallak, M.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States